CLINICAL TRIAL: NCT01594307
Title: Blood Pressure Monitor Clinical Test (Cuff Range: 13.5 Cm-22cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AndonHealth7
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-04

CONDITIONS: Blood Pressure
Keywords: BP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- blood pressure monitor: Cuff circumference:13.5cm-22cm
- stethoscopy: Cuff circumference: 13.5cm-22cm

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a preformed cuff ranged 13.5 cm-22 cm.

ELIGIBILITY:
Inclusion Criteria:

* cuff circumference: 13.5cm-22cm

Ages: 23 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: resident of a community
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2012-02; Study Completion 2012-04 (Actual)